CLINICAL TRIAL: NCT02863263
Title: A Pilot Study to Evaluate Efficacy and Safety of Hydrophilic Polyurethane Foam Dressing in Patients With Pressure Ulcer
Brief Title: Efficacy and Safety of MedifoamⓇ and BetafoamⓇ in Pressure Ulcer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in meeting recruitment target
Sponsor: Mundipharma Pte Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BTF16-AP-401
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Pressure Ulcer
Keywords: foam dressing; MedifoamⓇ; BetafoamⓇ; povidone iodine
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Foam Dressing (Other): Over the course of 12 weeks, dressing is performed twice weekly, but additional dressing changes are allowed, depending on the condition of the pressure ulcer such as excessive exudates on the ulcer. The frequency of dressing change is limited to once daily.
  Interventions: Device: Foam Dressing
- Foam Dressing with Povidone Iodine (Other): Over the course of 12 weeks, dressing is performed twice weekly, but additional dressing changes are allowed, depending on the condition of the pressure ulcer such as excessive exudates on the ulcer. The frequency of dressing change is limited to once daily.
  Interventions: Device: Foam Dressing with Povidone Iodine

INTERVENTIONS:
Device: Foam Dressing — The purpose of the study is not to compare between the 2 devices, but to determine the efficacy of each type of device on its own. Subjects are randomised to one of 2 arms.
  Other Names: Brand name: MedifoamⓇ
  Arms: Foam Dressing
Device: Foam Dressing with Povidone Iodine — The purpose of the study is not to compare between the 2 devices, but to determine the efficacy of each type of device own. Subjects are randomised to one of 2 arms.
  Other Names: Brand name: BetafoamⓇ
  Arms: Foam Dressing with Povidone Iodine

SUMMARY:
This study aims to exploratively assess the efficacy and safety of hydrophilic polyurethane foam dressing (MedifoamⓇ or BetafoamⓇ) in pressure ulcer specifically. The target enrolment is 20 patients, with 10 patients per arm.

DETAILED DESCRIPTION:
As the primary objective, the percentage of completely healed patients and the time to complete healing will be assessed after applying the study device, MedifoamⓇ or BetafoamⓇ, for 12 weeks to pressure ulcer patients. In addition, the pressure ulcer size reduction rate over 12 weeks will be evaluated.

Patients will make once weekly site visits. There are 14 visits in total, including a screening visit 14 days (maximum) before the baseline visit.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged at least 19 years old as of the consent date
2. Pressure ulcer of National Pressure Ulcer Advisory Panel (NPUAP) Stage III at screening
3. Pressure ulcer size of 3-10 cm2 at screening
4. Written consent provided by the subject or representative

Exclusion Criteria:

1. Any study ulcer of NPUAP Stage I, II or IV
2. Diabetic ulcer or venous ulcer (or stasis ulcer)
3. Past history of surgical treatment within 1 year or irradiation at the target pressure ulcer within 1 year
4. Hypersensitivity reaction to this product or povidone iodine
5. Hyperthyroidism or thyroid disorder requiring drug treatment
6. Signs of a current underlying systemic infection (sepsis/bacterial infection/tuberculosis) or cellulitis or osteomyelitis
7. Type 1 diabetes
8. Current malnutrition
9. Heavy smoker: Current smoking level of ≥1 pack (20 cigarettes)/day of tobacco
10. Drug or alcohol addiction
11. Requirement of immune-suppressants during the study, or current chemotherapy or radiotherapy
12. Application of other investigational product/medical device within 1 month prior to the investigational device application
13. Pregnant or breast-feeding women
14. Other renal, hepatic, neurological or immunological disorder that may interfere with the wound healing process, at the discretion of the Investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-07-29 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harsha Arumugam, Study Director — Mundipharma Singapore Holding Pte. Limited
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Foam Dressing | Foam Dressing With Povidone Iodine
Started | 3 | 2
Completed | 2 | 1
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Foam Dressing | Foam Dressing With Povidone Iodine | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Complete Healing of Ulcer Within 12 Weeks
Description: Complete healing is defined as epithelial tissue covering 100% of the ulcer, with intact dermis and epidermis and without abrasion or ulceration.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Foam Dressing | Foam Dressing With Povidone Iodine
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

2. Primary Outcome: Time to Complete Healing of Ulcer Within 12 Weeks as Measured by Number of Days From Baseline
Description: as for outcome 1
Time Frame: 12 weeks
Population: There is no analysis and result for this outcome measure as none of the subjects achieved complete healing of ulcer within 12 weeks.
Arm/Group | Foam Dressing | Foam Dressing With Povidone Iodine
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Pressure Ulcer Size Measured Using A Ruler at Week 12
Description: The ulcer area (for ulcers without re-epithelization) is measured at each visit after foam dressing application. A photograph of the ulcer is taken and a using a ruler (MediRuleⓇ) is used to measure its length and width to obtain the area in cm2.
Time Frame: Week 12 (Or Last Observation Carried Forward)
Population: Statistical analysis for this outcome measure was not performed due to low enrolment and early study termination.
Measure: Median (Full Range); unit: cm2
Arm/Group | Foam Dressing | Foam Dressing With Povidone Iodine
Number analyzed (Participants) | 3 | 2
cm2 | 5.05 [1.0 to 9.1] | 2.8 [0.5 to 5.1]

4. Secondary Outcome: Pressure Ulcer Scale for Healing (PUSH) Score Measured Using PUSH Tool Version 3.0 At Week 12
Description: The PUSH score is measured at alternate visits (2-week intervals) starting from baseline and will be compared against baseline.
  Minimum score= 0 Maximum score: 17 Higher score: worse outcome
Time Frame: Week 12 (Or Last Observation Carried Forward)
Population: Statistical analysis for this outcome measure was not performed due to low enrolment and early study termination.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Foam Dressing | Foam Dressing With Povidone Iodine
Number analyzed (Participants) | 3 | 2
score on a scale | 8 [5 to 11] | 7 [4 to 10]

5. Secondary Outcome: Number of Participants With a Dressing Change Frequency Greater Than Twice Per Week
Time Frame: 12 weeks
Population: The original Outcome Measure was frequency of additional dressing change. However, statistical analysis for this outcome measure was not performed due to low enrolment and early study termination. Therefore, the number of participants with dressing changes of more than twice weekly is reported instead.
Measure: Number; unit: participants
Arm/Group | Foam Dressing | Foam Dressing With Povidone Iodine
Number analyzed (Participants) | 3 | 2
participants | 3 | 2

6. Secondary Outcome: Number of Patients Achieving Early Study Completion Due to Complete Healing
Description: as for outcome 1
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Foam Dressing | Foam Dressing With Povidone Iodine
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With New Infections at the Pressure Ulcer Based on Clinical Signs and Symptoms Checklist (CCSC)
Description: Patients with at least 1 new infection after the foam dressing application at baseline until Visit 14 will be taken into account.
  Infection is defined as presence of purulent exudates or 2 or more symptoms stated in the CCSC. For patients with existing infection at baseline, infection is defined as the development of an additional symptom or recurrence of the baseline symptom after it was completely healed.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Foam Dressing | Foam Dressing With Povidone Iodine
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

8. Other Pre Specified Outcome: Safety as Evaluated by Number of Local Adverse Events at the Target Pressure Ulcer
Description: Examples of these local events are erythema, edema, itching, flare and rash.
Time Frame: 12 weeks
Measure: Number; unit: local adverse events
Arm/Group | Foam Dressing | Foam Dressing With Povidone Iodine
Number analyzed (Participants) | 3 | 2
local adverse events | 1 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Method of systematic assessment: Physical examination was done at every visit and laboratory test was done at the last visit.
Arm/Group | Foam Dressing | Foam Dressing With Povidone Iodine
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Foam Dressing (N=3) | Foam Dressing With Povidone Iodine (N=2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — The causal relationship was assessed to be unrelated to the investigational device.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Foam Dressing (N=3) | Foam Dressing With Povidone Iodine (N=2)
Pyrexia (General disorders) | 2 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pyuria (Infections and infestations) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Difficulties in meeting recruitment target led to termination of the trial. Statistical analysis was not performed due to insufficient number of subjects enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Mundipharma Pte Ltd is owner of the data. No Investigator may publish the results of this study without prior approval from Mundipharma Pte Ltd.

DOCUMENTS (2):
  • Study Protocol (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT02863263/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT02863263/SAP_001.pdf